CLINICAL TRIAL: NCT00879931
Title: Influence of Corticoids on Renal Function in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006/031
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Elective Cardiac Surgery
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): methylprednisolone
  Interventions: Drug: Methylprednisolone
- 2 (Placebo Comparator): Placebo (NaCl 0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone
  Arms: 1
Drug: Placebo — Placebo (NaCl 0.9%)
  Arms: 2

SUMMARY:
Hypothesis: Corticoid treatment in cardiac surgery works renal protective.

Study design: Randomized, double blind trial in which one group of patients will receive methylprednisolone and the other group (control) will receive placebo NaCl 0.9%.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-80 year
* patients scheduled for elective cardiac surgery.
* preoperative creatinine levels of < 2mg/dl
* no corticoid treatment

Exclusion Criteria:

* non-elective surgery
* patiënts with renal dysfunction: creatinine > 2mg/dl
* patiënts treated with corticoids

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Renal dysfunction and renal failure postoperatively in cardiac surgery | within 48 hours after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan Bouchez, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be